CLINICAL TRIAL: NCT02331706
Title: A Pilot Study to Determine the Feasibility of Conventional Induction Chemotherapy Followed by G-CSF Mobilized Donor Leukocyte Infusion (DLI) and IFN-α (IFN-DLI) for Relapsed Acute Leukemia After Allogeneic Stem Cell Transplantation.
Brief Title: IFN-DLI for Relapsed Acute Leukemia After Allo-SCT
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 09414
Record Dates: First submitted 2014-12-22; First posted 2015-01-06 (Estimated); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: Leukemia
MeSH Terms: conditions — Leukemia | interventions — Introns

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Subject Recipients (Experimental)
  Interventions: Drug: Interferon alpha-2B (IFN-α) 3 million units (MU) subcutaneous daily
- Subject Donors (Experimental)
  Interventions: Drug: Interferon alpha-2B (IFN-α) 3 million units (MU) subcutaneous daily

INTERVENTIONS:
Drug: Interferon alpha-2B (IFN-α) 3 million units (MU) subcutaneous daily

SUMMARY:
This trial is designed to determine the feasibility of conventional induction chemotherapy, IFNand G-CSF mobilized DLI (IFN-DLI) in subjects with relapsed AML and ALL after allo-SCT.

ELIGIBILITY:
Inclusion Criteria:

DLI Recipient

* Relapsed AML or ALL ≥ 60 days after allogeneic SCT.
* Evidence of residual donor chimerism on most recent analysis (within 4 weeks of enrollment).
* Age ≥ 18 years of age,
* Karnofsky performance status ≥ 60%.
* Absence of active GVHD and off immunosuppression. Subjects on tapering prednisone will be eligible if their dose is 0.25 mg/kg or less and being actively tapered. We suggest a 28 day waiting period off of immunosuppression but some subjects with rapidly progressive disease may need to be treated before 30 days and will still be eligible.
* Adequate organ function: Cr ≤ 2 mg/dL; ALT/AST < 3x ULN, direct bili <3x ULN.
* Matched sibling or un-related donor (A, B, C, and DR) available to undergo leukopheresis.
* Subjects must be able to sign consent and be willing and able to comply with scheduled visits, treatment plan and laboratory testing.
* Willing to provide blood samples for research purposes.
* Willing to adhere to medically accepted form of birth control to prevent pregnancy (includes: complete abstention from intercourse, condoms, diaphragms, cervical cap, intra-uterine device, history of surgical sterility - tubal ligation or vasectomy in patient or partner, or oral contraceptive).

DLI Donor

1. HLA identical to recipient subject.
2. Considered medically eligible for leukopheresis procedure by independent donor physician (University of Pennsylvania physician who is not the recipient's primary transplant physician for related donors; physician designated by National Marrow Donor Program for unrelated donors).
3. Considered medically eligible to receive G-CSF (filgrastim) by independent donor physician.

Exclusion Criteria

Recipient

* Prior cell therapy for relapse within the past 90 days.
* Requirement for active immunosuppression to treat GVHD.
* Pregnant or lactating women. The safety of this therapy on unborn children and effects on breast milk are not known.
* Uncontrolled active infection
* Any uncontrolled active medical disorder that would preclude participation as outlined.

Donor

- Unable to participate in a leukopheresis procedure or receive G-CSF (filgrastim).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2016-11-11 (Actual); Study Completion 2017-11-11 (Actual)

PRIMARY OUTCOMES:
Number of Adverse Events | 2 years

SECONDARY OUTCOMES:
overall survival | 2 years
disease-free survival | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: David Porter, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States